CLINICAL TRIAL: NCT00242489
Title: A Placebo-Controlled, Parallel-Group, Double-Blind Study to Assess Safety and to Define the Clinically Effective Dose Range of MK0663 in Patients With Osteoarthritis of the Knee, Followed by a Double-Blind, Active-Comparator-Controlled Extension.
Brief Title: Etoricoxib in the Treatment of Osteoarthritis (MK-0663-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-007; 2005_088
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Arcoxia
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib; Diclofenac

INTERVENTIONS:
Drug: MK0663, etoricoxib / Duration of Treatment: Part I (6 weeks), Part II (8 weeks)
Drug: Placebo;Diclofenac 50mg(tid)/Duration of Treatment: Part I (Placebo) 6 weeks;Part II (Diclofenac) 8 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of etoricoxib in the treatment of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years of age with a clinical diagnosis of Osteoarthritis (OA)of the knee for 6 months prior to study entry (ARA class I, II, or III).
* Positive therapeutic effect from prior NSAID therapy.
* Worsening of symptoms upon withdrawal of prior treatment.
* With the exception of OA, in otherwise good health

Exclusion Criteria:

* Weight no more than 280 pounds (male or female).
* Recent, sustained use of gastroprotective agents.
* History of arthroscopy of the affected knee within 6 months prior to study entry.
* History of acute ligamentous or meniscal injury of the study joint within the previous 2 years.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1167 (Actual)
Dates: Start 1998-06; Primary Completion 1999-02 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
WOMAC Pain Subscale, Investigator Global Assessment of Disease Status, and Patient Global Assessment of Response to Therapy (not a primary endpoint in extension periods)

SECONDARY OUTCOMES:
Physical Function Subscale (WOMAC), Stiffness Subscale (WOMAC), Patient Global Assessment of Disease Status, Investigator Global Assessment of Response to Therapy , Proportion of Patients Discontinued Due to Lack of Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Gottesdiener K, Schnitzer T, Fisher C, Bockow B, Markenson J, Ko A, DeTora L, Curtis S, Geissler L, Gertz BJ; Protocol 007 Study Group. Results of a randomized, dose-ranging trial of etoricoxib in patients with osteoarthritis. Rheumatology (Oxford). 2002 Sep;41(9):1052-61. doi: 10.1093/rheumatology/41.9.1052. PMID 12209041
- [Result] Curtis SP, Bockow B, Fisher C, Olaleye J, Compton A, Ko AT, Reicin AS. Etoricoxib in the treatment of osteoarthritis over 52-weeks: a double-blind, active-comparator controlled trial [NCT00242489]. BMC Musculoskelet Disord. 2005 Dec 1;6:58. doi: 10.1186/1471-2474-6-58. PMID 16321158